CLINICAL TRIAL: NCT05218694
Title: Coronary Computed Tomography Angiography For Optimized Invasive Coronary examInation
Acronym: CT-FOCI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aarhus University Hospital Skejby (Other)
Responsible Party: Principal Investigator, Nicolaj Brejnholt Støttrup, MD, Ph.D., Aarhus University Hospital Skejby
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CT-FOCI01
Record Dates: First submitted 2021-12-03; First posted 2022-02-01 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Ischemic Heart Disease; Coronary Artery Disease
Keywords: CCTA
MeSH Terms: conditions — Myocardial Ischemia; Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Patients (n=120) are randomized 1:1
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CT-guided algorithm (CTGA) (Experimental): In the CTGA group only the artery suspected of having obstructive coronary disease is examined. Anatomy of the vessel, optimal viewing projections and choice of catheter is determined. A guiding catheter is used as first choice based on the artery involved and the aortic anatomy. Time is recorded according to the ST group, with timepoint 1 after conclusion of the angiogram, timepoint 2 after FFR.
  Interventions: Diagnostic Test: CCTA guided focused coronary angiography examination.
- Standard treatment (ST) (No Intervention): ST includes the use of two diagnostic cathers and examination of both coronary arteries by at least 6 different standard projections best optimizing the view of the coronary lesions.
  Additional projections may be included if deemed necessary for optimal angiographic evaluation

INTERVENTIONS:
Diagnostic Test: CCTA guided focused coronary angiography examination. — Focused examination based on Images from CCTA, by choice of optimal catheter used and projection.
  Arms: CT-guided algorithm (CTGA)

SUMMARY:
Coronary computed tomography angiography (CCTA) is a non-invasive method for visualization of the coronary arteries. The anatomical information obtained by CCTA, however, is rarely integrated into a subsequent coronary intervention. The CT-FOCI trial aims to evaluate, in a randomized setting, the benefit of implementing the information obtained by CCTA as part of the invasive examination using a CT-guided algorithm (CTGA). Patients (n=120) with symptoms of stable angina pectoris will be randomized 1:1 after CCTA has determined at least 1 stenosis with luminal diameter reduction of minimum 50% in a vessel segment > 2 mm in diameter. Subsequent, invasive examination and intervention will utilize the information available according to randomization. Primary efficacy endpoints are a reduction in patient radiation exposure, procedure time, procedural utensils, and contrast use.

Secondary endpoints is significant stenosis in the non-target vessel, only available in the conventional group.

DETAILED DESCRIPTION:
The study is a randomized, single center trial. Patients (n=120) referred for CCTA due to symptoms suggesting obstructive coronary disease (shortness of breath on exertion or angina in relation to activity), are randomized 1:1 if CCTA finds coronary lesions suggestive of obstructive coronary artery disease in at lest one vessel and thus indication for further investigation by invasive examination.

The patients are randomized to a standard treatment (ST) and a protocol with a CT-guided algorithm (CTGA) for optimal interventional work-flow. ST includes the use of two diagnostic cathers and examination of both coronary arteries by at least 6 different standard projections best optimizing the view of the coronary lesions. Additional projections may be included if deemed necessary for optimal angiographic evaluation. Procedural time consumption (timepoint 1) is measured at the completion of the angiogram as specified (7.4.2). If there is a switch to a guiding catheter and subsequent coronary physiology test (fractional flow reserve [FFR]) this is marked at timepoint 2 at the conclusion of the FFR.

In the CTGA group only the artery suspected of having obstructive coronary disease is examined. Anatomy of the vessel, optimal viewing projections and choice of catheter is determined. A guiding catheter is used as first choice based on the artery involved and the aortic anatomy. Time is recorded according to the ST group, with timepoint 1 after conclusion of the angiogram, timepoint 2 after FFR.

On the day of invasive examination, the total amount of contrast, radiation dose, procedural time consumption and cost of utensils are registered as primary endpoints. In the conventional group, any significant stenosis in the non-target vessel

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 and < 81 years
* Stable angina
* at least 1 vessel disease in either the left coronary artery or right coronary artery
* Stenosis grater than 50% and no stenosis greater than 40% on contralateral vessel unless fractional flow reserve by CT (FFRct) >0.80
* Vessel segment > 2 mm in diameter
* Subject eligible for Dual Anti Platelet Therapy (DAPT

Exclusion Criteria:

* Significant bleeding risk or other contraindications against heparinization or DAPT
* Known pregnancy
* Life expectancy < 120 days
* Patient unable to provide informed consent
* Patients with CTO (Chronic Total Occlusion).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Patient radiation dose | Through angiography completion, an average of 4-5 minuets. Timepoint 1
  After coronary angiography and percutaneous coronary intervention (PCI), the Dose Area Product (DAP) Gycm2 and the radiation time (MM:SS) is recorded.
Procedure time | Through angiography completion, an average of 4-5 minuets. Timepoint 1
  The procedure time is defined at the time from first catheter insertion to final catheter removal. Time is recorded in MM:SS.
Contrast use | Through angiography completion, an average of 4-5 minuets. Timepoint 1
  The amount of contrast medium used for examination and intervention is measured (ml) by weight measurements (gram = ml).
utensils use | Through angiography completion, an average of 4-5 minuets. Timepoint 1
  The use of utensils are logged and a cost estimate subsequently calculated on the basis of the current price list (DKK/USD).

SECONDARY OUTCOMES:
Stenosis in non-target vessel | Through angiography completion, an average of 4-5 minuets. Timepoint 1
  Significant stenosis in non-target vessel, (only conventional grope), confirmed by FFR <0.80

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Depart. of Cardiology, Aarhus N, Central Region, Denmark

IPD SHARING:
Plan to Share IPD: No